CLINICAL TRIAL: NCT06233058
Title: A Bioequivalence Study of Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets Relative to Yasmin® in Healthy Thai Female Volunteers Under Fasting Condition
Brief Title: Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets Relative to Yasmin®
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bio-innova Co., Ltd (Industry)
Responsible Party: Principal Investigator, Sasitorn Kittivoravitkul, Principal Investigator, Bio-innova Co., Ltd
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DRE-027-22
Record Dates: First submitted 2023-12-15; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Healthy Subjects
Keywords: Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1-Drospirenone+ Ethinyl Estradiol test product and then reference product (Experimental): Participants will receive treatment 1 in period 1 and treatment 2 in period 2. Where treatment 1= Drospirenone 3 mg + Ethinyl Estradiol 0.03 mg Tablets test product, treatment 2= Drospirenone 3 mg + Ethinyl Estradiol 0.03 mg Tablets reference product.
  Interventions: Drug: Drospirenone+ Ethinyl Estradiol Tablets-Test product
- Sequence 1-Drospirenone+ Ethinyl Estradiol reference product and then test product (Experimental): Participants will receive treatment 2 in period 1 and treatment 1 in period 2. Where treatment 1= Drospirenone 3 mg + Ethinyl Estradiol 0.03 mg Tablets test product, treatment 2= Drospirenone 3 mg + Ethinyl Estradiol 0.03 mg Tablets reference product.
  Interventions: Drug: Drospirenone+ Ethinyl Estradiol Tablets-Reference product

INTERVENTIONS:
Drug: Drospirenone+ Ethinyl Estradiol Tablets-Test product — Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets Manufactured by: Umeda Company Limited, Thailand
  Arms: Sequence 1-Drospirenone+ Ethinyl Estradiol test product and then reference product
Drug: Drospirenone+ Ethinyl Estradiol Tablets-Reference product — Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets Manufactured by: Bayer AG, Berlin, Germany
  Arms: Sequence 1-Drospirenone+ Ethinyl Estradiol reference product and then test product

SUMMARY:
The study is to compare the rate and extent of absorption of a generic formulation with that of a reference for mulation when given as equal labeled dose. The study will be randomized, open-label, single dose, two way crossover design with two-period, two-treatment and two-sequence under fasting condition and at least 28 days washout period between the doses.

DETAILED DESCRIPTION:
Title A Bioequivalence study of a randomized, open-label, single dose, two-way crossover design with two-period, two-treatment and two-sequence of Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets relative to Yasmin® in healthy Thai female volunteers under fasting condition.

Objectives The primary objective is to compare the rate and extent of absorption of a generic formulation with that of a reference formulation when given as equal labeled dose. The secondary objective is to evaluate the safety after oral administration of both test and reference formulation in healthy Thai female volunteers.

Study Design Randomized, open-label, single dose, two-way crossover design with two-period, two-treatment and two-sequence under fasting condition and at least 28 days washout period between the doses.

Sample Size 32 Healthy Human Thai female subjects. Two extra subjects if available, may be checked-in on the day of check in of period-I to compensate for any dropout prior to dosing of period-I. These subjects will be dosed if there are dropouts prior to dosing in period-I. If there are no dropouts, these subjects will be checked-out without being dosed after completion of dosing in period-I.

Drug-Product Test-Product: Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets Reference-product: Yasmin® (Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets) Manufactured by: Bayer AG, Berlin, Germany

Administration After an overnight fasting at clinical facility of at least 10 hours, each volunteer will receive a single dose of two tablets of Drospirenone (3 mg) + Ethinyl Estradiol (0.03 mg) Tablets of either test or reference with 250 mL of drinking water. Each volunteer will be allowed to drink water as desire except 1 hour before and after drug administration. The formulation is given in a crossover fashion as per the randomization schedule. After the administration, the subject's oral cavity will be checked by using flashlight to confirm complete medication and fluid consumption by pharmacist.

Blood Schedule In each period, a total of 21 blood samples (approximately 10 mL each) will be collected pre-dose (0 hour) and at 0.333, 0.667, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 4.500, 6.000, 8.000, 12.000, 16.000, 24.000, 36.000, 48.000 and 72.000 hours after study drug administration, respectively. The sample collection at 36.000, 48.000 and 72.000 hours after dosing will be on ambulatory basis (i.e. on separate visit.).

Sample Collection Blood samples will be collected through an indwelling catheter placed in a vein using disposable syringe or through fresh venipuncture with disposable syringes and needles. Approximately 10 mL blood sample will be collected and transferred to 2 sample collection tubes containing K3EDTA as anticoagulant at each sampling time point. After collection of blood samples from all the subjects at each time point, samples will be centrifuged at 4000 rpm for 5 minutes at 4±2°C. After centrifugation, each sample collection tube will be distributed into pre-labeled 3 cryovials, approximately 1.5 mL of plasma will be divided equally into another 3 cryovials, 3 of each analysis will be set as original (O) and Duplicate (D), Triplicate (T) respectively. Thereafter, Cryovials containing plasma sample will be stored at -70±10 °C.

Analytical Method Drospirenone and Ethinyl Estradiol plasma concentration will be assayed as per international Guidelines/In-house SOP by using a UPLC-MS/MS method.

Pharmacokinetic Parameters Drospirenone Primary pharmacokinetic parameter: Cmax, AUC0→ 72 and secondary pharmacokinetic parameter: Tmax, T1/2, Kel will be determined from the plasma concentration data of analytes.

Ethinyl Estradiol Primary pharmacokinetic parameter: Cmax, AUC0→t, AUC0→∞ and secondary pharmacokinetic parameter: Tmax, T1/2, Kel, AUC % Extrap will be determined from the plasma concentration data of analytes.

Statistical Analysis Drospirenone ANOVA, two one-sided tests for bioequivalence, for log-transformed pharmacokinetic parameters Cmax, AUC0→72 will be performed.

Ethinyl Estradiol ANOVA, two one-sided tests for bioequivalence, for log-transformed pharmacokinetic parameters Cmax, AUC0→t, AUC0→∞ will be performed.

Acceptance Criteria for Bioequivalence Drospirenone To be considered as bioequivalent, the 90% CI of Cmax, AUC0→72 of Drospirenone of test and reference products should be in the interval of 80-125% for the log-transformed data Ethinyl Estradiol To be considered as bioequivalent, the 90% CI of Cmax, AUC0→t, AUC0→∞ of Ethinyl Estradiol of test and reference products should be in the interval of 80-125% for the log-transformed data.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to provide written informed consent prior to participate in the study.
2. Healthy Thai female subjects are between 18 to 55 years of age.
3. The Body Mass Index (BMI) ranges from 18.5 to 30 kg/m2.
4. Comprehensive of the nature and purpose of the study and compliance with the requirement of the entire protocol and allow investigators to draw 7 mL of blood for monitoring subjects' safety after the completion of the study.
5. Negative urine pregnancy test for women and no breast-feeding.
6. Absence of significant diseases or clinically significant abnormal laboratory values on the laboratory evaluations, medical history or surgery during the screening. Some of the laboratory values e.g. Complete blood count etc. that out of the normal range will be carefully considered by physician.

Exclusion Criteria:

1. History or evidence of allergy or hypersensitivity to Drospirenone or Ethinyl Estradiol or any related drugs or any of the excipients of this product.
2. Subject with B.P. is Systolic B.P <90, ≥140 mm/Hg, Diastolic B.P <60, ≥90 mm/Hg, pulse rate >100 beats per minute.
3. Serum bilirubin greater than 1.5 times the upper limit of reference range (ULRR).*
4. Serum creatinine greater than 1.5 times the upper limit of reference range (ULRR).*
5. Alanine amino transferase (ALT) or aspartate amino transferase (AST) greater than 2 times the upper limit of reference range (ULRR).*
6. Positive of hepatitis B or C virus.
7. Have more than one abnormal EKG, which is considered as clinically significant. *
8. History or evidence of heart (heart attack, angina pectoris), renal, hepatic disease, adrenal insufficiency, pulmonary obstructive disease, bronchial asthma, hypertension, vascular disease (deep vein thrombosis, pulmonary embolism, venous thromboembolism, stroke, transient ischemic attack), migraine with aura, diabetics with vascular complications, metabolic disorder, or glaucoma
9. History or Family history of VTE in a first degree relative under the age of 45.
10. History of abnormal vaginal bleeding or coagulopathy.
11. History or Family history in a first degree of breast cancer.
12. History or evidence of gastrointestinal disorder likely to influence drug absorption or previous GI surgery other than appendectomy.
13. Any major illness in the past 3 months or any significant ongoing chronic medical illness.
14. History of psychiatric disorder or depression
15. History of regular alcohol consumption exceeding 7 drinks/week for females (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of hard liquor) and cannot stop at least 2 days before the study drug administration and until the completion of each period of the study.
16. History of usually smoking (more than 10 cigarettes per day within past 1 year), if moderate smokers (less than 10 cigarettes per day) cannot stop at least 7 days before the study drug administration and until the completion of each period of the study.
17. High caffeine consumption (more than 5 cups of coffee or tea per day) and cannot stop at least 2 days before the study drug administration and until the completion of each period of the study.
18. History of pomelo or grapefruit or grapefruit products consumption and cannot stop at least 7 days before the study drug administration and until the completion of each period of the study.
19. History of St. John's Wort products consumption and cannot stop at least 28 days before the study drug administration and until the completion of the study.
20. Positive drug abused test in urine (Benzodiazepines, Marijuana (THC), Methamphetamine, Cocaine and Opioids).
21. Receipt of any prescription drug therapy within 14 days or 5 half-lives (whichever longer) preceding the first dose of study medication or over-the-counter (OTC) drugs or herbal medicines/food supplement within 7 days or hormonal methods of contraception within 28 days (Depo-Provera must be discontinued at least 6 months) prior to receiving the first dose of study medication.
22. History of difficulty in accessibility of veins in left and right arm.
23. Blood donation (one unit or 450 mL) within the past 3 months before the study.
24. Participation in any clinical study within the past 3 months before the study.
25. Subjects who are unwilling or unable to comply with the lifestyle guidelines described in this protocol.

(* Depend on decision of principal investigator and/or clinical investigator)

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2024-03-05 (Estimated); Primary Completion 2024-04-29 (Estimated); Study Completion 2024-05-27 (Estimated)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve from time zero to the last measurable concentration (AUC 0-t) | Blood samples will be collected for PK analyses in each period pre-dose (0 hour) and at 0.333, 0.667, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 4.500, 6.000, 8.000, 12.000, 16.000, 24.000, 36.000, 48.000 and 72.000 hours post-dose
  pre-dose (0 hour) and at 0.333, 0.667, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 4.500, 6.000, 8.000, 12.000, 16.000, 24.000, 36.000, 48.000 and 72.000 hours post-dose
Maximal measured plasma concentration (Cmax) | Blood samples will be collected for PK analyses in each period pre-dose (0 hour) and at 0.333, 0.667, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 4.500, 6.000, 8.000, 12.000, 16.000, 24.000, 36.000, 48.000 and 72.000 hours post-dose
  pre-dose (0 hour) and at 0.333, 0.667, 1.000, 1.333, 1.667, 2.000, 2.333, 2.667, 3.000, 3.500, 4.000, 4.500, 6.000, 8.000, 12.000, 16.000, 24.000, 36.000, 48.000 and 72.000 hours post-dose

SECONDARY OUTCOMES:
Number of subjects with adverse events | Approximately the day 28 after the last visit
  An adverse event (AE) is any untoward medical occurrence in a clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product

IPD SHARING:
Plan to Share IPD: No
No Company Policy